CLINICAL TRIAL: NCT03292601
Title: Effect of Feedback and Monitoring on Patient Compliance With Spinal Orthoses for Scoliosis Treatment
Brief Title: Brace Monitoring for Adolescent Idiopathic Scoliosis (AIS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AAAP4760
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Spinal Orthosis; Spinal Brace
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Intervention Model Description: (No Feedback Group was removed in 2019)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Feedback Group (Experimental): Participants will receive the standard-of-care scoliosis brace fitted with the compliance-monitoring study device and/or a temperature monitor (Orthotimer or iButton). The physician or a member of the research team will explain how the study device works to the patient and her/his parent. The physician or member of the research team will also explain the feedback mechanisms that exist to inform the patient that s/he has fit the device to the clinician-indicated appropriate tension and the online component of the program that allows for brace tension monitoring.
  Interventions: Device: NYRC Brace Scoliosis Monitor

INTERVENTIONS:
Device: NYRC Brace Scoliosis Monitor — Scoliosis Monitor is a system that allows the continuous monitoring of the scoliosis brace use compliance and posture. This product includes a brace wearable that enables the monitoring of the scoliosis brace. The wearable device is able to communicate with a companion mobile application which stores and processes the collected data and is responsible for data synchronization.
  Other Names: Monitor

SUMMARY:
The overall aim of the study is to utilize a novel device and smartphone application in order to improve measurement of patient compliance with at-home bracing for scoliosis as well as create a more accurate assessment of brace fit via continuous and objective measures of tension. These ground-breaking metrics will provide analyzable data to more accurately reflect and predict actual patient compliance as well as allow for further exploration of how to increase compliance, and thus, efficacy of bracing; it will additionally allow both physicians and patients to have a more reliable measure for brace fit by providing them with continuous data of fit via tension, and provide built-in feedback mechanisms to the patient to ensure proper tightness of the brace.

Additionally, the study will investigate whether providing the wearer's own brace-wear compliance information directly to the patient and their caregiver(s) via the mobile app will further improve rates of compliance as compared to those who do not receive the same feedback mechanism.

DETAILED DESCRIPTION:
The current method to set brace tension is subjective; it is limited to the attending clinician making a mark on the brace straps, to which the patient tightens the straps during daily wear. Once the strap is set in place, the current standard-of-care does not involve any more monitoring. Therefore, ideal strap tension is unknown and the effectiveness of bracing may be unknowingly compromised by many as yet unidentified variables. In recent years, a small number of studies have emerged related to the strap tension of bracing yet no clear guidelines on correct strap tension currently exist. Considering the potential effects on preventing scoliosis progression and brace-associated complications, the need for guidelines regarding optimal brace fit are greatly needed for clinical use. Via this brace monitoring study, continuous monitoring of tension at brace fitting, throughout the day, and related to positional changes will be possible with a very minimal device and smartphone application. The tremendous amounts of data generated by the device and its app will be used to create a database from which our team will gather information about brace wear compliance and use tension information for the development of standards for effective strap tension associated with greater scoliosis curve correction. Lastly, the effect of a patient's engagement with his or her brace - through the smartphone app - will be examined. It is well established in the literature that observation increases compliance, but no studies investigating patient self-monitoring through personal devices currently exists. This is a vital area of investigation given the recent explosion in personal health-assessing devices e.g. the Apple watch, Up band, fitbit, etc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Adolescent Idiopathic Scoliosis (AIS)
* Sanders skeletal stage 4 or earlier
* Clinician-recommended Rigo bracing
* Patient receiving brace treatment

Exclusion Criteria:

- Prior spine surgery

Ages: 8 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Wear Time Compliance | Up to 1 year
  Measured as number of hours that the patient actually wore the brace.
Wear Compliance: Valid Hours | Up to 1 year
  Measured as time (in hours) that the brace was worn to the provider-prescribed tightness
In-Brace Curve Correction Rate | Up to 1 year
  In-brace curve correction will be analyzed by an in-brace radiograph to determine the degree of immediate curve correction (absolute change in degrees).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Roye, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital of NY Presbyterian/Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided